CLINICAL TRIAL: NCT02134730
Title: School-based Universal Prevention for Anxiety and Depression in Sweden: A Cluster-randomized Trial Using the FRIENDS for Life Manual
Brief Title: School-based Universal Prevention for Anxiety and Depression in Sweden: A Cluster-randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AGJA-01
Record Dates: First submitted 2014-04-15; First posted 2014-05-09 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Anxiety Disorders
Keywords: FRIENDS for life; universal prevention; school children; anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wait list (No Intervention): Schools in waitlist condition will be offered the intervention after the 12-months follow up. Waitlist means that the schools work as usual with issues of mental health.
- FRIENDS for life (Experimental): The intervention is delivered for 10 consecutive weeks, 60 minutes per session.
  Interventions: Behavioral: FRIENDS for life

INTERVENTIONS:
Behavioral: FRIENDS for life — Friends for life (FFL). The FFL is a prevention program created by professor Paula Barrett, Brisbane, Australia. It is based on cognitive behavioral treatment strategies, for example the link between thoughts and feelings, negative and positive thoughts, breathing and relaxing exercises, support from others, breaking challenging situation in smaller steps, and problem-solving techniques. The children's workbook comprises practice-sheets for use during class, and homework assignments. The group leader manual comprises detailed instructions to all exercises.
  Arms: FRIENDS for life

SUMMARY:
Mental illness is a major health problem in children and young people, and there is evidence that mental illness is increasing among young people in the population. More than 80 % of the cost to society of mental illness in children in Sweden is the cost of treatment and care.

Anxiety and depression are the most common psychiatric problems in children and adolescents.

In comparison with the treatment of mental disorders, there is relatively limited knowledge about prevention. There are at least two very important reasons to investigate further preventive interventions for anxiety and depression. (1) Only about 20% of children and adolescents with anxiety or depression use health services. (2) Some children stop treatment and almost 40% do still fulfill criteria for the disorder after treatment.

FRIENDS for life is one of the most evaluated prevention programs internationally. The program has shown promising results in research. The overall aim of the present study is to evaluate FRIENDS for Life in Sweden.

DETAILED DESCRIPTION:
Mental illness is a major health problem in children and young people, and there is evidence that mental illness is increasing among young people in the population. More than 80 % of the cost to society of mental illness in children in Sweden is the cost of treatment and care. Only a small portion thus consists of preventive interventions. The report "Programs to prevent mental illness in children - a systematic literature review" (2010) from the Swedish National Council on Technology Assessment (SBU), concluded that no prevention program has evidence of efficacy under Swedish conditions. A target for future prevention work is according to the authors SBU-report that programs that are used have scientific support and evaluated in Sweden. Based on the review the report's authors recommend that five programs should be prioritized for further evaluation. One of these five programs is FRIENDS for life, a prevention program to prevent anxiety.

Anxiety and depression are the most common psychiatric problems in children and adolescents. Untreated anxiety disorders often have a chronic course or may occur again and depression in adolescents often continue into adulthood anxiety and depression in children and adolescents predicts a variety of psychiatric diagnoses later in life, leading to difficulties with school and friends, and lead to increased risk of suicidal acts, alcohol and drug abuse.

In comparison with the treatment of mental disorders, there is relatively limited knowledge about prevention. There are at least two very important reasons to investigate further preventive interventions for anxiety and depression. (1) Only about 20% of children and adolescents with anxiety or depression use health services. (2) Some children stop treatment and almost 40% do still fulfill criteria for the disorder after treatment.

FRIENDS for life is one of the most evaluated prevention programs internationally. The program has shown promising results in research. In Sweden there are no high-quality evaluation of prevention programs targeting anxiety and depression. Based on the high incidence of anxiety and depression and its serious consequences it is of utmost importance to investigate whether prevention programs work in a Swedish context. The overall aim of the present study is to evaluate FRIENDS for Life in Sweden. The following research questions guide the study:

1. Do FRIEND for life affect children's estimates of anxiety and depression symptoms and parents' estimates of children's anxiety symptoms, on the scales Spence Children's Anxiety Scale? Is the possible impact still visible after 12 months?
2. Do FRIEND for life affect the presence of anxiety diagnoses and subclinical anxiety at 12 months according to ADIS-C/P interview?

   Additional research questions are:
3. Is there any congruence between parents' and children's estimates of the child's anxiety symptoms?
4. Do FRIEND for life affect parents' and teachers' estimates of children's general mental health?
5. Do gender, symptom level, fidelity to the manual, decreased negative thoughts, behavioral inhibition affect the effect of FRIEND for life?

International studies have shown promising results of FRIEND for life. Previous studies have, however, been of varying quality. Strengths of this study are that parents, teachers and children are respondents, and it is investigated whether various background characteristics and implementation factors influence the effect.

Given the high prevalence of anxiety and depression in young ages, and the fact that only a few children with anxiety and depression use health services, the knowledge that this study generates are very important.

ELIGIBILITY:
Inclusion Criteria:

* Written parental consent

Exclusion Criteria:

* No other exclusion criteria since of universal prevention

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 695 (Actual)
Dates: Start 2013-09; Primary Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in SCAS (Spence Children's Anxiety Scale) | Participants are assessed pre intervention, post intervention and up to 12-months
  Additional assessments using a short version of the SCAS (12 items out of 44) are made at two occasions during intervention (october and november 2013)

SECONDARY OUTCOMES:
The Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID) | Assessed up to 12-months
Change in Children's Depression Inventory (CDI) | Assessed pre intervention, post intervention and up to 12 months
Change in Strengths and Difficulties Questionnaire (SDQ) | Assessed pre intervention, post intervention and up to 12 months follow-up
  SDQ is rated by participants' parents and teachers

CONTACTS AND LOCATIONS:
Overall Officials: Ata Ghaderi, Dr., Principal Investigator — Karolinska Institutet
Locations (1):
- Department of Psychology, Uppsala University, Uppsala, Sweden